CLINICAL TRIAL: NCT06382818
Title: Personalization of Breast Radiotherapy According to Loco-regional Recurrence Risk and Toxicity Probability
Acronym: PROBA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2023-10 PRO
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Radiotherapy breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: * COHORT A = Low risk of recurrence / Low risk of breast toxicity
  * COHORT B = Low risk of recurrence / High risk of breast toxicity
  * COHORT C = High risk of recurrence / Low risk of breast toxicity
  * COHORT D = High risk of recurrence / High risk of breast toxicity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COHORT A (Other): In this cohort, the patients with low risk of recurrence and a low risk of breast toxicity
  Interventions: Radiation: COHORT A
- COHORT B (Other): For this cohort, patients with low risk of recurrence and a high risk of breast toxicity, will receive breast radiotherapy according to the investigator's decision among:
  * External partial : 40 Gy in 15 fractions to the partial breast only (tumorectomy bed).
  * Exclusive Brachytherapy: 30.1 Gy in 7 fractions or 32.0 Gy in 8 fractions of high-dose-rate brachytherapy in 5 days or as 50 Gy of pulsed-dose-rate brachytherapy over 5 treatment days.
  * Whole Breast Normo fractionated with Fixed Field Intensity Modulated radiotherapy(IMRT) Technique: 50 Gy in 25 daily fractions over 5 weeks +/- Sequential (+ 16 Gy/8fr) or SIB (simultaneous integrated boost) (60 Gy/25 fr) treatment for boost if applicable.
  Interventions: Radiation: COHORT B
- COHORT C (Other): For this cohort, patients with high risk of recurrence and a low risk of breast toxicity, will receive whole breast and nodes Hypofractionated VMAT and a localized simultaneous boost according to the HypoG01 schema protocol:
  VMAT Technique, 42.3 Gy in 18 fractions on all target volume on 3.5 weeks +/- SIB boost if need (52.2Gy in 18 fractions).
  Interventions: Radiation: COHORT C
- COHORT D (Other): For this cohort, patients with high risk of recurrence and a high risk of breast toxicity, will receive breast radiotherapy based on available clinical trials:
  - Whole Breast and Nodes Hypofractionated VMAT with adaptive treatment (margin reduction): HypoG01 Schema with VMAT Technique, 42.3 Gy in 18 fractions on all target volume over 3.5 weeks +/- SIB boost if need (52.2Gy in 18 fr) In case of patient refusal or technique unavailable, a standard treatment available in the center for this indication will be delivered.
  Interventions: Radiation: COHORT D

INTERVENTIONS:
Radiation: COHORT A — IMRT radiotherapy on whole breast according to the investigator's decision among:
  * Moderate whole breast hypofractionated RT according to the START B schema with Fixed Field IMRT Technique: 40.05 Gy in 15 daily fractions over 3 weeks and a Sequential boost (+ 16 Gy/8 fr) or (+13.5/5 fr) if applicable.
  * Extreme whole breast hypofractionated RT according to :
    * The FAST schema: Once-a-week ultra-HypoRT with Fixed Field IMRT Technique, 28.5 Gy in 5 fractions in 5 weeks
    * The FAST-Forward schema: Very accelerated course of HypoRT with Fixed Field IMRT Technique, 26 Gy in 5 fractions in 5 consecutive days
  Arms: COHORT A
Radiation: COHORT B — Breast radiotherapy according to the investigator's decision among:
  * External partial VMAT: 40 Gy in 15 fractions to the partial breast only (tumorectomy bed).
  * Exclusive Brachytherapy: 30.1 Gy in 7 fractions or 32.0 Gy in 8 fractions of high-dose-rate brachytherapy in 5 days or as 50 Gy of pulsed-dose-rate brachytherapy over 5 treatment days.
  * Whole Breast Normo fractionated IMRT with Fixed Field IMRT Technique: 50 Gy in 25 daily fractions over 5 weeks +/- Sequential (+ 16 Gy/8fr) or SIB (60 Gy/25 fr) treatment for boost if applicable.
  Arms: COHORT B
Radiation: COHORT C — Whole breast and nodes Hypofractionated VMAT and a localized simultaneous boost according to the HypoG01 schema protocol:
  VMAT Technique, 42.3 Gy in 18 fractions on all target volume on 3.5 weeks +/- SIB boost if need (52.2Gy in 18 fractions).
  Arms: COHORT C
Radiation: COHORT D — Breast radiotherapy based on available clinical trials:
  - Whole Breast and Nodes Hypofractionated VMAT with adaptive treatment (margin reduction): HypoG01 Schema with VMAT Technique, 42.3 Gy in 18 fractions on all target volume over 3.5 weeks +/- SIB boost if need (52.2Gy in 18 fr) In case of patient refusal or technique unavailable, a standard treatment available in the center for this indication will be delivered.
  Arms: COHORT D

SUMMARY:
Our objective is based on a personalized approach of adjuvant breast radiotherapy by selecting patients according to tumor recurrence and toxicity risk.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women in the world and remains a major public health burden with 25% of all cancer cases and 15% of all cancer deaths among females. The Incidence has increased with the introduction of mammography screening and continues to rise, mainly due to population aging; meanwhile, breast cancer survival has significantly improved over the past decades.

Adjuvant radiotherapy (RT) is an essential component of the treatment. After breast surgery for invasive carcinoma, RT is commonly used and delivered without considering the different tumor subtypes, unless the node involvement risk, because it decreases the rate of local recurrence and by this way, specific mortality. The " one size fits all " approach is widely applied, with two main options: breast or chest wall only radiotherapy or breast or chest wall plus nodes radiotherapy. Rare are the centers that discuss IMRT use, external partial breast irradiation, adaptive breast necessity, etc….

1. Breast cancer and loco-regional recurrence risk Ten-year cancer specific survival exceeds 70%, with 89% survival for local and 62% for regional disease. The risk of recurrence is high during the first two years after the initial diagnosis for patients with hormonal receptor (HR)-negative breast cancer, but rapidly decreases below the recurrence risk of HR-positive tumors.

   Loco-regional recurrence (LRR) occurs in 5-15% of cases treated with breast conservative surgery (BCS) plus adjuvant radiotherapy (RT) or mastectomy and is considered an independent poor prognostic factor6. The management of LRR requires a multidisciplinary approach. Total mastectomy is the standard of care for isolated LRR after BCS. However, secondary BCS ± RT is an alternative approach that could be discussed case by case.

   Parameters to predict the risk of recurrence are those included in the NHS UK updated PREDICT score such as age, node status, tumor grade, proliferation index, Her2 and hormone receptor expression.
2. Adjuvant breast radiotherapy and subcutaneous toxicity probability Severe but also moderate toxicities after curative-intent radiotherapy (RT), such as fibrosis, retraction or telangiectasia with poor cosmetic outcome can have a negative impact on quality of life following breast cancer and a marked effect on subsequent psychological outcome. Multiple factors are known to increase the risk of radiation toxicity including individual radiosensitivity9. While the toxicity risks for patients are well-established, determining an individual's normal tissue radiosensitivity is rarely possible before treatment.

   Nevertheless, current practice standards often prescribe radiation dose and volume without regard to individual radiosensitivity.

   In that context, a normal tissue radiosensitivity test that includes a rapid (72h) radiosensitivity assay based on flow cytometric assessment of radiation-induced CD8 (cytotoxic T cells 8) T-lymphocyte apoptosis (RILA) was developed by Ozsahin et al. A prospective study was conducted to determine whether the RILA assay could help identifying patients at high risk of severe toxicities. The RILA assay was performed in 399 patients with different cancer types before RT. Findings confirmed that patients who developed severe toxicities displayed a compromised apoptotic response.

   More recently, the RILA assay was validated in a prospective multicenter trial with more than 500 patients with breast cancer. The negative predictive value for grade ≥2 breast fibrosis was 91% for RILA scores ≥20% and the positive predictive value was 22% for RILA scores <12% (the overall prevalence of grade ≥2 breast fibrosis was estimated at 14%). For the first time, RILA as a continuous variable was significantly associated with toxicities. Recently, the French results have been validated by a prospective European trial with similar predictive values of the RILA.

   In the CO-HO-RT trial, the RILA assay was used as the main stratification factor and no late toxicity occurred in patients with a RILA score >16%.

   In 2022, the RILA assay was included in the French recommendation (RECORAD) as the only validated predictive test for post-radiotherapy toxicity in a large, multi-center, prospective study.

   Based on these data, the NovaGray RILA Breast® test has been developed and combine both a biological analysis (radio-induced lymphocyte apoptosis) and an algorithmic analysis.

   The NovaGray RILA Breast is an vitro diagnostic medical device (IVMD) pertaining CE-mark. This prognostic test that assesses the risk of developing grade 2+ breast fibrosis at 36 months following radiotherapy. The test is performed on a blood draw and results are provided within a week, which does not delay the beginning of the radiotherapy.
3. Matrix approach according to tumor recurrence and toxicity risk When using a predictive radiosensitivity test in clinical practice, an alternative treatment must be available to the patient in case of an unfavourable result, i.e. an adjustment in the radiotherapy protocol (change in fractionation or total dose), the addition or elimination of a concomitant treatment (e.g. chemotherapy) or the absolute contraindication to radiotherapy in highly radiosensitive patients for whom the treatment-related risk may be greater than the expected benefit.

Based on tumor control probability (TCP) and normal tissue complication probability (NTCP) we can group the patients into four situations described below.

1. Clinical situation #1 : High TCP(Tissue Complication Probability) / Low NTCP (Normal Tissue Complication Probability) : COHORT A This circumstance is the optimum situation: a high local control probability and a low risk of developing toxicity. In this situation, the total dose of radiotherapy could be limited to the strict necessity since the probability of tumor control is already high. However, alternative fractionations such as moderate hypofractionated can be proposed to shorten the duration of treatment. In breast cancer, a regimen delivering 42.5 Gy in 16 fractions or 40 Gy in 15 fractions can be offered according to the Canadian or UK (united kingdom) regimen,. Recently, hypofractionated regimen are becoming more extreme with shorten fractionation regimen over 5 weeks or over 1 week . From a radiobiological and economic standpoint, these short regimens can provide a benefit in terms of quality of life with a lower cost of treatment.

   All of them are now included in the recommendations of the French National Society of Radiation Oncology and the French National Cancer Institute (INCa, Cancers du sein - Recommendations et outils d'aide à la pratique (e-cancer.fr)). All are considered as an option in daily clinical practice.
2. Clinical situation #2 : High TCP / High NTCP : COHORT B In this situation, the patient is at risk of developing toxicity, but the probability of tumor control is high). In those cases, possible alternatives to radiotherapy may be discussed such as surgical treatment alone. In breast cancer, this can mean offering total mastectomy for a small tumor (possibly with immediate breast reconstruction) to postpone the indication of adjuvant radiotherapy. For a tumor with a very favorable prognosis, namely after 65 years old, avoiding radiotherapy after breast surgery may also be an option. In that case, treatment with partial irradiation of the breast (using external technique or brachytherapy) can also be proposed, to improve the long-term cosmetic results, while ensuring good local control.

   All of them are now included in the recommendations of the French National Society of Radiation Oncology. All are considered as an option in daily clinical practice.
3. Clinical situation #3 : Low TCP / Low NTCP : COHORT C In that situation, the patient is at low risk of developing toxicity but the probability of tumor control is low. One of the possibilities is to increase the total dose of radiotherapy, namely with a localized boost within the tumor bed in invasive disease 5 and nodes irradiation according to the HypoG trial.

   This treatment is also included in the recommendations of the French National Society of Radiation Oncology.
4. Clinical situation #4 : Low TCP / High NTCP : COHORT D This is the most unfavourable situation, with a radiation-resistant tumor and a patient with a high risk of developing toxicity. Dose de-escalation cannot be proposed to decrease toxicity in such cases, as the risk of tumor recurrence may be too high. Alternative fractionations, such as hyperfractionation (moderate or high depending on the organs at risk) could however be useful by decreasing the risk of toxicity while retaining a satisfactory level of tumor control. These regimens have not been validated and discussions should be carried out on a case-by-case basis. However, the impact on the decrease of toxicity, especially late-onset toxicity, has yet to be demonstrated. If adjusted radiotherapy regimens are not feasible and standard oncological treatment administered, the radioprotection of normal tissue should be discussed using adaptive techniques as it could decrease the risk of toxicity while maintaining good tumor control.

In this specific COHORT, inclusion in a new clinical trial evaluating adaptive treatment will be proposed to the patient. In case of patient refusal or technique unavailable, a standard treatment available in the center for this indication will be delivered.

ELIGIBILITY:
Inclusion Criteria:

General criteria (for all cohorts):

1. Women ≥ 18 years old.
2. Invasive breast cancer treated by conservative or radical surgery.
3. Conservative breast cancer surgery or radical mastectomy.
4. Indication of breast irradiation.
5. Extension evaluation of disease will be proven negative (M0).
6. Negative pregnancy test (blood or urine at the choice of investigator), to be carried out within 7 days of registration, for women of childbearing age only.
7. Effective contraception for women of childbearing age
8. Must be geographically accessible for follow-up.
9. Written and dated informed consent.
10. Affiliated to the French national social security system.

    Cohort A and B:

    - Low risk of recurrence (all of the criteria)

    • pT1-T2
    * SBR (Scarff Bloom et Richardson grade) grade ≤ 2 (low grade)
    * ER+ and / or PR+ (hormone-receptor positive)
    * cN0/pN-
    * HER 2 -
    * Ki67 ≤10%

    pN- with T3-4 and grade 3 and internal tumor will be considered at high risk of recurrence and will be proposed node irradiation (and will be switched to COHORT C or D).

    Cohort C and D:

    - High risk of recurrence (pN+ and at least one of all) adapted from the UK PREDICT

    • ER- and PR-

    • HER2 amplified

    • pT3-4

    • SBR grade ≥ 3
    * KI67 > 10%

    Cohort A and C:
    * Low risk of breast toxicities identified by the NovaGray RILA Breast® test

    Cohort B and D:

    - High risk of breast toxicities identified by the NovaGray RILA Breast® test

    Exclusion Criteria:
    * 1. Patients with distant metastases.

2. Patients with breast DCIS (ductal carcinoma in situ) 3. Concomitant bilateral breast cancer 4. Previous breast radiotherapy 5. Patients with previous or concomitant other (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years.

6. Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.

7. Patients known to be HIV positive (no specific tests are required to determine the eligibility).

8. Patients known as hypersensitive to radiation 9. Patients treated with systemic investigational drugs during the present study (Observational cohorts are accepted if the collection of data does not interfere with the current trial) 10. Pregnant or breast-feeding women 11. Patient unable to comply with study obligations for geographic, social, or physical reasons, or who is unable to understand the purpose and procedures of the study 12. Person deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 854 (Estimated)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2028-03-06 (Estimated); Study Completion 2038-03-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients without any grade 2 or more fibrosis, nor radio-induced sarcoma | at 10 years
  Toxicity free survival is defined as the interval between date of inclusion and the occurrence of fibrosis grade 2 or more or radio-induced sarcoma. Patients without event at the analysis will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Acute toxicity | from the start of RT to 12 weeks post RT
  according to NCI-CTCAE v5 is defined as side effects observed
Late toxicity | from 12 weeks post RT to 3, 5 and 10 years post RT
  according to NCI-CTCAE v5 is defined as side effects observed
Local recurrence rate (LRR) | at 3, 5, 10 years
  LRR will be deducted from the local recurrence survival defined as the interval between date of inclusion and the occurrence of local relapse. Patients without local relapse at the analysis will be censored at the date of last follow-up
Relapse-free survival (RFS) rate | at 3, 5, 10 years
  RFS is defined as the interval between date of inclusion and the occurrence of relapse. Patients without relapse at the analysis will be censored at the date of last follow-up
Overall survival (OS) rate | at 3, 5, 10 years:
  OS is defined as the interval between date of inclusion and the occurrence of death, due to any cause. Patients alive at the analysis will be censored at the date of last follow-up.
Radiation-induced Breast Sarcoma prevalence | at 10 years
  Prevalence of Radio-induced Breast Sarcoma at 10 years will be estimated using the Kaplan-Meier method, and then described using rate at 10 years with its associated 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: AZRIA DAVID, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Institut Du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No